CLINICAL TRIAL: NCT07060313
Title: TARGETING DUAL PATHWAYS IN REFRACTORY COCCYDYNIA: A COMPARATIVE STUDY OF GANGLION IMPAR BLOCK ALONE VERSUS COMBINED WITH PERICOCCYGEAL INJECTION
Brief Title: TARGETING DUAL PATHWAYS IN REFRACTORY COCCYDYNIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mert Zure, Mert Zure, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Health Sciences University
Record Dates: First submitted 2025-07-08; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Coccydynia
Keywords: Coccydynia; Spinal Injections; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: A standard procedure was applied to all patients by the same pain medicine specialist with over 5 years of experience, in a sterile operating room under fluoroscopic guidance and monitored conditions. The patients underwent noninvasive blood pressure monitoring, pulse oximetry, and a five-lead electrocardiogram [ECG], and intravenous access was established in the forearm before positioning for the intervention. The position used during the intervention was the prone position, with a pillow placed under the belly. The procedure area was disinfected with povidone-iodine and covered with a sterile drape. Anterior-posterior (AP) imaging was first performed with a C-arm scopy device, which was then placed in the lateral position.
  The ganglion impar was accessed with a Quincke spinal needle, transsacrococcygeally (from between the first and second coccygeal vertebrae if sacrococcygeal access could not be achieved). Then, 1 mL of non-ionic contrast medium was administered, and fluoroscopic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ganglion Impar Block Group (Active Comparator): This group of participants received ganglion impar block only.
  Interventions: Procedure: Ganglion Impar Block
- Combination Therapy Group (Active Comparator): This group of participants underwent pericoccygeal injection in addition to impar block.
  Interventions: Procedure: Ganglion Impar Block and Pericoccygeal Injection

INTERVENTIONS:
Procedure: Ganglion Impar Block — The ganglion impar was accessed with a Quincke spinal needle, transsacrococcygeally (from between the first and second coccygeal vertebrae if sacrococcygeal access could not be achieved). Then, 1 mL of non-ionic contrast medium was administered, and fluoroscopic anterior-posterior and lateral imaging was performed to confirm the appropriate spread of contrast (Figure 1). After this confirmation, 2 mL of 0.5% bupivacaine, 2 mL of saline, and 40 mg of methylprednisolone acetate were injected.
  Arms: Ganglion Impar Block Group
Procedure: Ganglion Impar Block and Pericoccygeal Injection — In the combination therapy group who underwent pericoccygeal injection in addition to impar block, following the same procedure, 5 mL of 0.25% bupivacaine and 20 mg of methylprednisolone were injected into the posterior pericoccygeal region while the needle was withdrawn, thus also targeting blockade of the anococcygeal nerve.
  Arms: Combination Therapy Group

SUMMARY:
This retrospective cohort study included 60 patients aged 18-65 years treated at a tertiary pain clinic between June 2022 and June 2024. Patients received either Ganglion Impar Block (GIB) alone or GIB combined with pericoccygeal injection in a single session under fluoroscopic guidance. Pain severity and functional outcomes were assessed using the Numeric Rating Scale (NRS-11), Oswestry Disability Index (ODI), and Paris Functional Coccydynia Impact Questionnaire (PFCIQ) before the procedure and at 1 and 3 months post-intervention.

DETAILED DESCRIPTION:
Study Design and Population This retrospective study compared the effects of GIB alone versus GIB combined with pericoccygeal injection in coccydynia patients treated at the Pain Clinic of Kanuni Sultan Süleyman Training and Research Hospital. The study cohort was drawn from patients with a confirmed diagnosis of coccydynia persistent for at least 3 months as determined by history, clinical examination, and radiological imaging, who had undergone either GIB or GIB with pericoccygeal injection, and had complete medical records available for review between June 2022 and June 2024. Patients having a recent intervention (in the past 6 months), morbid obesity (BMI > 35 kg/m²), severe comorbidities, skin infections, bleeding disorders, pregnancy, or having incomplete records were excluded. A total of 60 patients aged 18-65 years who underwent either GIB or GIB with pericoccygeal injection were included. The sample size was determined using a power analysis (effect size: 0.84, power: 80%, error margin: 5%), based on previously published studies reporting significant differences in pain and functional outcomes following ganglion impar block interventions. Accordingly, a minimum of 30 patients per group was required, and a total of 60 patients were enrolled.

Intervention A standard procedure was applied to all patients by the same pain medicine specialist with over 5 years of experience, in a sterile operating room under fluoroscopic guidance and monitored conditions. The patients underwent noninvasive blood pressure monitoring, pulse oximetry, and a five-lead electrocardiogram [ECG], and intravenous access was established in the forearm before positioning for the intervention. The position used during the intervention was the prone position, with a pillow placed under the belly. The procedure area was disinfected with povidone-iodine and covered with a sterile drape. Anterior-posterior (AP) imaging was first performed with a C-arm scopy device, which was then placed in the lateral position.

The ganglion impar was accessed with a Quincke spinal needle, transsacrococcygeally (from between the first and second coccygeal vertebrae if sacrococcygeal access could not be achieved). Then, 1 mL of non-ionic contrast medium was administered, and fluoroscopic anterior-posterior and lateral imaging was performed to confirm the appropriate spread of contrast. After this confirmation, 2 mL of 0.5% bupivacaine, 2 mL of saline, and 40 mg of methylprednisolone acetate were injected.

In the combination therapy group who underwent pericoccygeal injection in addition to impar block, following the same procedure, 5 mL of 0.25% bupivacaine and 20 mg of methylprednisolone were injected into the posterior pericoccygeal region while the needle was withdrawn, thus also targeting blockade of the anococcygeal nerve.

After the procedure, all patients were monitored and observed for at least two hours. Patients who had no additional complaints during follow-up visits were discharged.

Data Collection Data were extracted from patient files following ethical approval. Recorded information included demographic details (age, sex), body mass index (BMI), symptom duration, comorbidities, prior medical treatments, procedure details, coccydynia etiology, and outcome measures.

Outcome Measures Pain Assessment with the Numeric Rating Scale (NRS-11) Pain levels were measured using the Numeric Rating Scale (NRS-11), a widely recognized tool for quantifying pain intensity. This scale ranges from 0 to 10, where 0 represents no pain and 10 signifies the worst imaginable pain. Patients were asked to rate their pain based on their subjective experience, providing a straightforward and reliable metric for assessing pain severity. The NRS-11 was administered before the procedure and at follow-up intervals of 1 and 3 months post-procedure to track changes in pain levels over time, allowing for a clear evaluation of the intervention's effectiveness in reducing pain.

Oswestry Disability Index (ODI) Functional disability was assessed using the Oswestry Disability Index (ODI), a validated questionnaire designed to evaluate the impact of pain on daily functioning. The ODI consists of 10 domains-pain intensity, lifting, self-care, walking, sitting, sexual function, standing, social life, sleep quality, and travel-each scored on a 0-5 scale. The total score is expressed as a percentage (0-100%), with higher scores indicating greater disability. This comprehensive tool captures the multidimensional impact of pain on patients' lives . ODI scores were collected pre-procedure and at 1 and 3 months post-procedure to monitor improvements in functional capacity following the intervention.

The Paris Functional Coccydynia Impact Questionnaire (PFCIQ) To specifically address coccyx-related functional limitations, the Paris Functional Coccydynia Impact Questionnaire (PFCIQ) was employed. This targeted questionnaire evaluates the unique challenges associated with coccydynia, including difficulties with sitting, standing, or performing activities that exacerbate coccyx pain. The PFCIQ provides a detailed assessment of how coccyx-specific impairments affect patients' quality of life and daily activities. Like the other metrics, PFCIQ scores were recorded before the procedure and at 1 and 3 months post-procedure, enabling a focused evaluation of the intervention's impact on coccyx-related functional outcomes.

Ethical Considerations The study was approved by the institutional ethics committee of Kanuni Sultan Süleyman Training and Research Hospital on 26/09/2024 (ID: KAEK/2024.09.200). As it is a retrospective cohort study, no additional patient consent beyond routine clinical consent was required. Data collection occurred between October 1, 2024, and December 1, 2024.

ELIGIBILITY:
Inclusion Criteria:

* with a confirmed diagnosis of coccydynia persistent for at least 3 months as determined by history, clinical examination, and radiological imaging, who had undergone either GIB or GIB with pericoccygeal injection, and had complete medical records available for review between June 2022 and June 2024.

Exclusion Criteria:

* having a recent intervention (in the past 6 months), morbid obesity (BMI > 35 kg/m²), severe comorbidities, skin infections, bleeding disorders, pregnancy, or having incomplete records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Pain Assessment with Numeric Rating Scale 11 | From the beginning of the treatment to the 3 month follow-up
  Pain levels were measured using the Numeric Rating Scale (NRS-11), a widely recognized tool for quantifying pain intensity. This scale ranges from 0 to 10, where 0 represents no pain and 10 signifies the worst imaginable pain. Patients were asked to rate their pain based on their subjective experience, providing a straightforward and reliable metric for assessing pain severity. The NRS-11 was administered before the procedure and at follow-up intervals of 1 and 3 months post-procedure to track changes in pain levels over time, allowing for a clear evaluation of the intervention's effectiveness in reducing pain.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | From the beginning of the treatment to the 3 month follow-up
  Functional disability was assessed using the Oswestry Disability Index (ODI), a validated questionnaire designed to evaluate the impact of pain on daily functioning. The ODI consists of 10 domains-pain intensity, lifting, self-care, walking, sitting, sexual function, standing, social life, sleep quality, and travel-each scored on a 0-5 scale. The total score is expressed as a percentage (0-100%), with higher scores indicating greater disability. This comprehensive tool captures the multidimensional impact of pain on patients' lives. ODI scores were collected pre-procedure and at 1 and 3 months post-procedure to monitor improvements in functional capacity following the intervention.
The Paris Functional Coccydynia Impact Questionnaire (PFCIQ) | From the beginning of the treatment to the 3 month follow-up
  To specifically address coccyx-related functional limitations, the Paris Functional Coccydynia Impact Questionnaire (PFCIQ) was employed. This targeted questionnaire evaluates the unique challenges associated with coccydynia, including difficulties with sitting, standing, or performing activities that exacerbate coccyx pain. The PFCIQ provides a detailed assessment of how coccyx-specific impairments affect patients' quality of life and daily activities. Like the other metrics, PFCIQ scores were recorded before the procedure and at 1 and 3 months post-procedure, enabling a focused evaluation of the intervention's impact on coccyx-related functional outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Istanbul Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Genc Perdecioglu GR, Yildiz G. Coccygeal Nerve Blockade vs. Impar Ganglion Blockade in Coccydynia: A Randomised Clinical Trial. Cureus. 2024 Sep 10;16(9):e69118. doi: 10.7759/cureus.69118. eCollection 2024 Sep. PMID 39398734
- [Background] Sencan S, Yolcu G, Bilim S, Kenis-Coskun O, Gunduz OH. Comparison of treatment outcomes in chronic coccygodynia patients treated with ganglion impar blockade versus caudal epidural steroid injection: a prospective randomized comparison study. Korean J Pain. 2022 Jan 1;35(1):106-113. doi: 10.3344/kjp.2022.35.1.106. PMID 34966017